CLINICAL TRIAL: NCT03840291
Title: Resolution of Thrombi in Left Atrial Appendage With Edoxaban
Acronym: REFLEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Daiichi Sankyo Korea Co., Ltd., a Daiichi Sankyo Company (Industry)
Responsible Party: Principal Investigator, Seongwook Han, Professor of Internal Medicine, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-09-041
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Thrombosis
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edoxaban treatment (Experimental): 1. Men or women aged ≥ 20 years with NVAF patients who has LAA thrombi documented by transesophageal echocardiography (TEE) up to 72 hours prior to start of study medication are eligible.
  2. Patients in this group are taking Lixiana® (Edoxaban) 60mg for resolution of left atrial appendage thrombi
  3. Reduced (30mg) dose is administered in patients with one or more of the following clinical factors:
     * Moderate or severe renal impairment (creatinine clearance (CrCL) 15 - 50 mL/min)
     * Low body weight ≤ 60 kg
     * Concomitant use of the following P-glycoprotein (P-gp) inhibitors: ciclosporin,dronedarone, erythromycin, or ketoconazole.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Edoxaban will be used for resolution of left atrial appendage thrombi
  Other Names: Lixiana®

SUMMARY:
Non-valvular (NV) atrial fibrillation (AF) increases the risk of stroke by approximately fivefold. The atrial thrombi associated with AF are seen within the left atrial appendage (LAA) in most cases (> 90%). Anticoagulation with a vitamin-K antagonist (VKA) is recommended to prevent thromboembolic complications and to resolve thrombi. Non-VKA oral anticoagulants (NOACs) have replaced the VKA for the thromboprophylaxis in patients with NVAF since 2010. Therefore, NOAC can be the excellent alternative to VKA concerning resolving preexisting LAA thrombi because of its rapid onset of action and no need of bridging with heparin. However, there is still lack of data regarding the optimal treatment for patients with AF and thrombi in LAA with NOAC. There are only several case reports of the efficacy of NOACs in resolving LAA thrombi available.

Edoxaban, which has data showing efficacy and safety in thromboprophylaxis, can be the new option for treatment of patients with AF and LAA thrombi. The purpose of this study is to evaluate the efficacy of Edoxaban in resolving the LAA thrombi, which is related with nonvalvular AF.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 20 years
* Hemodynamically stable nonvalvular AF or atrial flutter
* LAA thrombus documented by TEE up to 72 hours prior to start of study medication
* VKA or NOAC-naïve or untreated within 1 month prior to sign the informed consent
* VKA pretreated but under the therapeutic International Normalized ratio levels (<2.0; documented with at least 2 consecutive measurements that are at least 24 hours apart) within last 6 weeks
* Women of childbearing potential and men must agree to use adequate contraception when sexually active

Exclusion Criteria:

* Transient Ischemic Attack within 3 days prior to study inclusion
* Severe, disabling stroke (modified Rankin score of 4-5, inclusive) within 3 months or any stroke within 14 days before the start of study drug
* Acute thromboembolic events or thrombosis (venous/arterial) within the last 14 days prior to study inclusion
* Acute myocardial infarction within the last 14 days prior to study inclusion
* Cardiac-related criteria: Previous intracardiac thrombus, Free-floating ball thrombus, Intracardiac tumor, known left ventricular or aortic thrombus
* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
complete resolution of LAA thrombi | 6 weeks
  The percentage of subjects with complete resolution of LAA thrombi

SECONDARY OUTCOMES:
Treatment responses of thrombi | 6 weeks
  Treatment responses of thrombi: Number of participants with resolved, reduced, unchanged, enlarged thrombi or newly appeared thrombi
Ischemic stroke event | 12 weeks
  The percentage of subjects who experienced ischemic stroke
Bleeding event | 12 weeks
  The percentage of subjects who experienced bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Seongwook Han, M.D., Ph.D., Study Chair — Keimyung University Dongsan Medical Center
Locations (12):
- South Korea (12):
  - Keimyung University Dongsan Medical Center, Daegu
  - Division of Cardiology, Department of Internal Medicine, Kyungpook National University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Yeungnam University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Daegu Catholic University Medical Center, Daegu
  - Catholic University of Korea, Incheon St. Mary's hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Cardiovascular Hospital, Seoul
  - Seoul Samsung Medical Center, Seoul
  - Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju